CLINICAL TRIAL: NCT00002550
Title: A Phase III Comparison Between Concurrent Chemotherapy Plus Radiotherapy and Concurrent Chemotherapy Plus Radiotherapy Followed by Surgical Resection for Stage IIIA (N2) Non-Small Cell Lung Cancer
Brief Title: Chemotherapy Plus Radiation Therapy With or Without Surgery in Treating Patients With Stage IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network); North Central Cancer Treatment Group (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9309; CDR0000063333; CAN-NCIC-BR13; CLB-9592; E-R9309; NCCTG-R9309; NCI-94-C-0043; SWOG-9336; INT-0139
Record Dates: First submitted 1999-11-01; First posted 2003-04-10 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT + chemotherapy followed by surgery + chemotherapy (Experimental): Induction radiation therapy (RT) + concurrent induction chemotherapy followed by surgery and additional chemotherapy
  Interventions: Drug: cisplatin; Drug: etoposide; Procedure: conventional surgery; Radiation: radiation therapy
- RT + chemotherapy followed by chemotherapy + RT (Active Comparator): Induction RT + concurrent induction chemotherapy followed by additional chemotherapy + RT
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Procedure: conventional surgery
  Arms: RT + chemotherapy followed by surgery + chemotherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells. It is not yet known if chemotherapy plus radiation therapy is more effective with or without surgery for lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combining cisplatin, etoposide, and radiation therapy with or without surgery in treating patients who have stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival, median (2-year) survival, and long-term (5-year) survival in patients with newly diagnosed, stage IIIA (N2) non-small cell lung cancer treated with radiotherapy concurrently with cisplatin and etoposide with or without surgical resection.

Secondary

* Compare the patterns of local and distant failure in patients treated with these regimens.
* Determine the relationship of tobacco use, alcohol use, and diet with toxicity of these regimens and outcome in both men and women.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by contralateral mediastinal sampling or biopsy (yes vs no), tumor stage (T1 vs T2 vs T3), and performance status (70-80% vs 90-100%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive induction with cisplatin IV over 1 hour on days 1 and 8 and etoposide IV over 1 hour on days 1-5. Treatment continues every 4 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning within 24 hours of the first dose of chemotherapy, patients undergo induction radiotherapy 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity. Patients without local progression or distant metastases at 2-4 weeks after completion of course 2 undergo resection approximately 3-5 weeks after completion of course 2. All visible, accessible bronchopulmonary, hilar, and mediastinal lymph nodes are excised. The choice of surgical procedure (thoracotomy, lobectomy, or pneumonectomy with en bloc resection of tumor extending into the parietal pleura, chest wall, pericardium, or diaphragm) is at the discretion of the surgeon. Patients who undergo resection receive 2 additional courses of chemotherapy alone beginning 4-6 weeks postoperatively. Patients with unresectable disease or who are medically unfit for or refuse resection receive 2 additional courses of chemotherapy alone beginning immediately after completion of course 2.
* Arm II: Patients undergo induction chemoradiotherapy as in arm I but do not undergo resection. Patients without local progression or distant metastases within 1 week before anticipated completion of induction radiotherapy receive 2 additional courses of chemotherapy beginning immediately after completion of course 2. Patients without local or distant progression after completion of course 4 undergo boost radiotherapy for 8 days.

Patients are followed every 2 months for 1 year, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 510 patients will be accrued for this study within 4.9 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven newly diagnosed, stage IIIA (T1-3, N2) non-small cell lung cancer

  * Eligible subtypes:

    * Adenocarcinoma
    * Large cell carcinoma
    * Squamous cell carcinoma
    * Nonlobar and nondiffuse bronchoalveolar cell carcinoma
* Measurable or evaluable disease on chest x-ray and/or contrast CT scan

  * Contrast thoracic CT required to complete staging
* Single primary bronchogenic tumor (no more than 1 parenchymal lung lesion)
* Pleural effusions allowed if 1 of the following conditions is met:

  * Negative cytology on thoracentesis if effusions present before mediastinoscopy or exploratory thoracotomy
  * Effusion seen on CT scan but not on chest x-ray and deemed too small to tap under CT or ultrasound guidance
* Positive ipsilateral mediastinal node(s) with or without positive ipsilateral hilar nodes

  * Mediastinal nodes separate from primary lesion on CT scan or surgical exploration
  * Histologic or cytologic proof of N2 disease by thoracotomy, mediastinoscopy, mediastinotomy, Chamberlain procedure, Wang needle, or fine needle aspiration under bronchoscopic or CT guidance
  * Nodal biopsy or aspiration waived if all of the following conditions are met:

    * Paralyzed left true vocal cord documented by bronchoscopy or indirect laryngoscopy
    * Nodes visible in Level 5 region on CT scan
    * Distinct primary lesion separate from nodes on CT scan
  * All mediastinal nodal involvement mapped (positive or negative)
* No positive nodes in contralateral mediastinum (supraclavicular areas and higher) and neck

  * Mediastinoscopy, mediastinotomy, Chamberlain procedure, or thoracotomy required for nodes larger than 1 cm on contrast CT scan
  * Surgery waived if nodes negative or no larger than 1 cm on CT scan
* Lymphadenopathy allowed if biopsy proof of a benign cause
* No metastases by contrast CT or MRI scan of the brain, bone scan, CT scan of the lungs to exclude other ipsilateral or contralateral parenchymal lesions, and contrast CT scan of the upper abdomen including entire liver and adrenals
* No hepatomegaly or splenomegaly by physical examination or CT scan unless documentation of a benign cause
* No pericardial effusion
* No superior vena cava syndrome
* No prior diagnosis of lung cancer

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 90-100% (70-80% allowed if albumin at least 0.85 times lower limit of normal and weight loss no greater than 10% within 3 months before diagnosis)

Hematopoietic:

* White blood cell count (WBC) at least 4,000/mm^3 OR
* Granulocyte count at least 2,000/mm^3
* Platelet count normal
* Hemoglobin at least 10.0 g/dL (less than 8.5 g/dL allowed if no marrow involvement with tumor)

Hepatic:

* See Performance status
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)*
* Serum glutamate oxaloacetate transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) no greater than 1.5 times ULN* NOTE: * Unless documentation of a benign cause

Renal:

* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No myocardial infarction within the past 3 months
* No active angina
* No unstable arrhythmia
* No congestive heart failure

Pulmonary:

* Forced expiratory volume at one second (FEV1) at least 2.0 liters OR
* Predicted postresection FEV1 at least 800 mL based on quantitative V/Q scan
* Diffusion capacity of lung for carbon monoxide (DLCO) at least 50% predicted (corrected for hemoglobin) if pneumonectomy planned or likely after induction chemotherapy

Other:

* No clinically significant hearing loss unless willing to accept the potential of further loss
* No symptomatic peripheral neuropathy
* No peptic ulcer disease under active treatment
* No other medical illness not controllable by appropriate medical therapy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or ductal or lobular carcinoma in situ of the breast
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent colony-stimulating factors

Chemotherapy:

* No prior chemotherapy for lung cancer
* No concurrent chemotherapy for another condition (such as arthritis)

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for lung cancer

Surgery:

* See Disease Characteristics
* No prior resection of primary tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 1994-03; Primary Completion 2004-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Median overall survival | From randomization to date of death or last follow-up. Analysis occurs after patients have been potentially followed for 2.5 years.

SECONDARY OUTCOMES:
Median Progression-free survival | From randomization to date of death or last follow-up. Analysis occurs after patients have been potentially followed for 2.5 years.
Patterns of local and distant failure | From randomization to date of failure (local, regional or distant progression). Analysis occurs after patients have been potentially followed for 2.5 years.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Ettinger, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Kathy S. Albain, MD, Principal Investigator — Loyola University; David H. Johnson, MD, Study Chair — Vanderbilt-Ingram Cancer Center; Bruce E. Johnson, MD, Study Chair — Dana-Farber Cancer Institute; Mark R. Green, MD, Study Chair — Medical University of South Carolina; Robert C. Miller, MD, Study Chair — Mayo Clinic; Yvon Cormier, MD, Study Chair — L'Hopital Laval
Locations (16):
- United States (15):
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - University of Rochester Cancer Center, Rochester, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CCOP - Green Bay, Green Bay, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Background] Machtay M, Bae K, Movsas B, Paulus R, Gore EM, Komaki R, Albain K, Sause WT, Curran WJ. Higher biologically effective dose of radiotherapy is associated with improved outcomes for locally advanced non-small cell lung carcinoma treated with chemoradiation: an analysis of the Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):425-34. doi: 10.1016/j.ijrobp.2010.09.004. Epub 2010 Oct 25. PMID 20980108
- [Background] Machtay M, Swann S, Komaki R, et al.: What is the meaning of local-regional control after chemoradiation for locally advanced NSCLC? An RTOG analysis. [Abstract] Lung Cancer 50 (Suppl 2): A-O-041, S17, 2005.
- [Result] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Result] Albain KS, Swann RS, Rusch VR, et al.: Phase III study of concurrent chemotherapy and radiotherapy (CT/RT) vs CT/RT followed by surgical resection for stage IIIA(pN2) non-small cell lung cancer (NSCLC): outcomes update of North American Intergroup 0139 (RTOG 9309). [Abstract] J Clin Oncol 23 (Suppl 16): A-7014, 624s, 2005.
- [Result] Albain KS, Scott CB, Rusch VR, et al.: Phase III comparison of concurrent chemotherapy plus radiotherapy (CT/RT) and CT/RT followed by surgical resection for stage IIIA(pN2) non-small cell lung cancer (NSCLC): initial results from intergroup trial 0139 (RTOG 93-09) . [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2497, 2003.
- [Result] Turrisi AT, Scott CB, Rusch VR, et al.: Randomized trial of chemoradiotherapy to 61 Gy [no S] versus chemoradiotherapy to 45 Gy followed by surgery [S] using cisplatin etoposide in stage IIIa non-small cell lung cancer (NSCLC): intergroup trial 0139, RTOG (9309). [Abstract] Int J Radiat Oncol Biol Phys 57 (2 Suppl): S125-6, 2003.